CLINICAL TRIAL: NCT02159131
Title: An Open-label Study to Evaluate the Pharmacokinetics of an Oral Contraceptive Containing Levonorgestrel and Ethinyl Estradiol When Co-administered With GSK1265744 in Healthy Adult Female Subjects
Brief Title: Study to Evaluate the Pharmacokinetics of an Oral Contraceptive Containing Levonorgestrel and Ethinyl Estradiol When Co-administered With GSK1265744 in Healthy Adult Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 117011
Record Dates: First submitted 2014-05-15; First posted 2014-06-09 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2014-12

CONDITIONS: Infections, Human Immunodeficiency Virus and Hepatitis
Keywords: ethinyl estradiol; GSK1265744; pharmacokinetics; oral contraceptive; oral contraceptive containing levonorgestrel and ethinyl estradiol; levonorgestrel
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; Hepatitis | interventions — Levonorgestrel; cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OC containing levonorgestrel and ethinyl estradiol + GSK126574 (Experimental): Eligible subjects will enter a run-in-period of 21 days (may extend to 49 days) to stabilize on OC containing levonorgestrel and ethinyl estradiol in order to synchronize the menstrual cycles of multiple subjects. Subjects completing run-in-period will enter Treatment period 1 and will be dosed OC once daily on Days 1 to 10. At day 11 subjects will enter Treatment period 2 and will be dosed with OC containing levonorgestrel and ethinyl estradiol + 744 once daily on Day 12 to 19. Subjects completing Treatment period 2 will have 7 OC free days (Day 22 to 28) during which withdrawal menses should occur. Subjects will then be followed up for 7 to 14 days (Day 28 to 35/49).
  Interventions: Drug: Ethinyl Estadiol; Drug: Levonorgestrel; Drug: GSK1265744

INTERVENTIONS:
Drug: Ethinyl Estadiol — EE is available as a combination of EE 0.03 mg and LNG 0.15mg, a monophasic oral contraceptive tablet to be taken along with 240 mL water
Drug: Levonorgestrel — LNG is available as a combination of EE 0.03 mg and LNG 0.15mg, a monophasic oral contraceptive tablet to be taken along with 240 mL water
Drug: GSK1265744 — GSK1265744 is available as 30 mg tablet to be taken along with 240 mL water

SUMMARY:
This open-label, fixed-sequence crossover study aims to evaluate the effect of GSK1265744 (744) oral administration on the pharmacokinetics (PK) and pharmacodynamics (PD) of a commonly used oral contraceptive (OC) product (combination of ethinyl estradiol and levonorgestrel), in 20 healthy female subjects. Each subject will participate in a Run-in Period (if needed), followed by a single-sequence Treatment Period. Subjects will receive oral contraceptive containing Levonorgestrel and Ethinyl Estradiol on Days 1 to 21 and be OC free on Days 22 to 28, during which withdrawal menses should occur. Subjects will receive OC alone on Days 1 to 10. Levonorgestrel (LNG) and ethinyl estradiol (EE) PK will be determined on Day 10. Subjects will then co-administer 744 and OC on Days 11 to 21. Levonorgestrel and ethinyl estradiol PK will be determined again on Day 21 to assess if co-administration with 744 results in a significant change in OC exposure compared to OC alone. Subjects will return to the study center for final follow-up evaluations 7 to 14 days after the last dose of study medication (Days 28 to 35).

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects, as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Females aged between 18 and 45 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Child-bearing potential with negative pregnancy test as determined by serum hCG test at screening AND agrees to use one of the contraception methods listed in the protocol in addition to OC (containing levonorgestrel and ethinyl estradiol ) from Day 1 of the Run-In Period (if required) or Day 1 of Treatment Period 1 until 14 days after the last dose of study drug to sufficiently minimize the risk of pregnancy. Female subjects must agree to use an additional form of contraception throughout the study and for the subsequent post-study follow-up period OR Has only same-sex partners, when this is her preferred and usual lifestyle.
* Female subject's with a body mass index (BMI) of 18to 30 kilogram per meter square (kg/m^2) and body weight >=50 kg (110 pounds [lbs]) and <114 kg (<250 lbs).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Alanine transaminase (ALT), alkaline phosphatase and bilirubin <=1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* History of any condition that would contraindicate OC administration (which may include hypertension, stroke, ischemic heart disease, venous thromboembolism or family history of thromboembolism, known factor V Leiden mutation or other gene mutations associated with increased risk of thromboembolism, migraine headaches, carcinoma of the breast, liver or endometrium, gallbladder disease, history of undiagnosed abnormal uterine bleeding, etc.).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 units for females. One unit is equivalent to 8 grams of alcohol: a half-pint (~240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* A positive pre-study Hepatitis B surface antigen (or positive Hepatitis B core antibody with negative hepatitis B surface antibody) or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen.
* A positive test for Human immunodeficiency virus (HIV) antibody.
* The subject's systolic blood pressure is outside the range of 80-140 millimeter of mercury (mmHg), or diastolic blood pressure is outside the range of 45-90mmHg.
* Exclusion criteria for screening ECG (Heart rate: <50 and >100 beats per minute [bpm], PR Interval: <120 and >220 milliseconds [msec], QRS duration: <70 and >120 msec, QTc interval [Bazett]: >450 msec): evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization); any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome); sinus pauses > 3 seconds; any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject; non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Women of childbearing potential who are unwilling or unable to use an appropriate method of contraception (see inclusion criteria) from at least Day 1 of the Run-in Period (if needed) or Day 1 of Treatment Period 1 until 14 days after the last dose of 744.
* Current or recent (within 6 months) users of tobacco-containing products.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Plasma (AUC[0-tau]) | Period 1: Predose on Day 9 and on Day 10: predose, and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose. Period 2: Predose on Day 20 and on Day 21 predose, and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose
  Blood samples will be collected to estimate the area under the concentration-time curve over the dosing interval (AUC[0-tau]) of LNG and EE following OC with and without 744

SECONDARY OUTCOMES:
Safety and tolerability of 744 when given with and without OC as assessed by adverse events (AE) | Up to 72 days
  Safety and tolerability as assessed by number of participants with AEs
Safety and tolerability of 744 when given with and without OC as assessed by clinical laboratory tests | Up to 72 days
  Safety laboratory parameters included hematology and clinical chemistry analysis and ECG
Safety and tolerability of 744 when given with and without OC as assessed by Electrocardiogram (ECG) | Up to 72 days
Safety and tolerability of 744 when given with and without OC as assessed by vital signs | Up to 72 days
  Vital signs will include pulse rate and blood pressure measurements
Composite of plasma pharmacokinetic (PK) parameters of 744 | Period 1: Predose on Day 9 and on Day 10: predose, and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose. Period 2: Predose on Day 20 and on Day 21 predose, and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose
  Maximum observed plasma concentration (Cmax), plasma concentration at the end of the dosing interval (Ctau), time to maximum drug concentration (tmax), and oral clearance (CL/F) CL/F will be used to evaluate the pharmacokinetics of LNG and EE after OC alone and after OC with 744.
Predose serum levels of Progesterone, Luteinizing hormone (LH) and follicle stimulating hormone (FSH) | At Screening and predose on Days 1, 10, 11, 21, and 22
  To assess the impact of 744 on the pharmacodynamic effects of OC on endogenous LH, FSH, and progesterone levels when given in combination compared with these parameters when OC is administered alone
Composite of plasma PK parameters of 744 - AUC(0-tau), Cmax, tmax, Ctau and CL/F | Predose on Day 20 and on Day 21: predose and at 1, 2, 3, 4, 6, 8, 12, and 24 hours post dose on Day 22
  To evaluate the PK of 744 when co-administered with LNG and EE

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, London, United Kingdom